CLINICAL TRIAL: NCT07295288
Title: Investigating the Efficacy of Botox Injections in Non-Cranial Nerve VII Innervated Muscles for Facial Synkinesis Management
Brief Title: Botox Injections in Non-Cranial Nerve VII Innervated Muscles for Facial Synkinesis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Priyesh Patel, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 251490
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Synkinesis
Keywords: botulinum toxin
MeSH Terms: conditions — Synkinesis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: The study design is a prospective crossover study. Patients who meet eligibility criteria and wish to proceed with the study will be randomized into two groups based on their MRN numbers. Patients with MRNs ending in an even number will undergo their standard BT injections (CN7 muscle groups only) + non-CN7 muscle groups at their first treatment session, followed by standard BT injections alone at their second treatment session. Patients with MRNs that end in an odd number will undergo the reverse injection process (standard BT injections alone at first treatment session, followed by standard BT injections + non-CN7 muscle groups at their second treatment session).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Even MRN (Other): Patients with MRNs ending in an even number will undergo their standard BT injections (CN7 muscle groups only) + non-CN7 muscle groups at their first treatment session, followed by standard BT injections alone at their second treatment session.
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]
- Odd MRN (Other): Patients with MRNs that end in an odd number will undergo the reverse injection process (standard BT injections alone at first treatment session, followed by standard BT injections + non-CN7 muscle groups at their second treatment session).
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [Botox] — Patients will receive standard of care synkinesis treatment. Depending on the treatment arm, they will receive additional botox injections to temporalis and masseter muscle groups which will only be injected on the ipsilateral side to the facial nerve injury. Decision to include the temporalis and/or masseter muscles will be based on each patients response to screening questions regarding jaw pain/tightness or headaches.

SUMMARY:
Facial synkinesis is a condition that occurs following facial nerve (CN7) injury, typically secondary to Bell's palsy, trauma, surgery (e.g., acoustic neuroma resection), or malignancy. Synkinesis is due to aberrant regeneration of the facial nerve, where axons regrow improperly and result in misdirected innervation of facial muscles. This results in involuntary, uncoordinated muscle movements, where activation of one muscle group triggers unintended contractions in others. Standard treatment of facial synkinesis involves botulinum toxin (BT) injections into muscles controlled by CN7 to reduce these unwanted movements. However, patients often anecdotally report that adding BT injections into non-CN7 innervated muscle groups, such as the masseter and temporalis muscles, improve their synkinesis symptoms. This study therefore aims to assess whether adding BT injections to non-CN7 innervated muscle groups, specifically the masseter and temporalis muscle, can improve treatment outcomes for people with facial synkinesis. This study will use a crossover design, where each participant will serve as their own control to compare treatment effects. In the first treatment arm, patients will receive only their standard BT injections into muscle groups controlled by CN7 - no other muscles will be treated. In the second treatment arm, will receive the same standard BT injections in CN7 muscles, plus additional injections into masseter and temporalis muscles. Patients will be randomized to a specific treatment arm at their first visit. At their second visit, they will be randomized to the other treatment arm, in standard crossover study design. Pre- and post-treatment surveys will be collected to assess the benefit of adding non-CN7 muscle groups.

DETAILED DESCRIPTION:
Facial synkinesis is a debilitating condition that occurs following injury to the facial nerve (CN7). It results from misdirected nerve regrowth, leading to involuntary, often conflicting muscle movements (e.g., eye closure during smiling or neck muscle tightening). This causes functional impairments (e.g., cheek biting, eating difficulties, reduced visibility), cosmetic concerns, and increased rates of anxiety and depression. Facial synkinesis has been reported in the literature to affect up to 75% of patients with facial nerve injury.

Chemodenervation of facial muscle groups using targeted BT injections has become a mainstay treatment for facial synkinesis. Typically, BT is selectively injected into hyperfunctioning CN7-innervated muscles on the injured side to allow for relaxation and restoration of organized muscle contraction. BT may also be injected into CN7-innervated muscles on the contralateral non-affected side, to improve facial symmetry. These injections have been shown across numerous studies to be safe, improve facial symmetry, and decrease severity of synkinesis symptoms. Injections are typically preformed every 3-6 months, depending on the needs of the patient and duration of injection benefit.

While synkinesis is thought to predominantly affect CN7 innervated muscles, in our clinical experience many patients also experience painful contracture of non-CN7 innervated muscles, such as the temporalis or master muscles. We therefore routinely inject these muscle groups with BT during patients synkinesis treatments. While patients anecdotally report that injection of non-CN7 innervated muscles improve their synkinesis symptoms in our clinical practice, this has not been systematically studied in the literature. This study therefore aims to investigate whether extending BT injections to non-cranial nerve 7-innervated muscles, specifically the masseter and temporalis muscle, can enhance outcomes for facial synkinesis.

Since participants are already receiving BT as standard care, the study introduces no additional risks, focusing only on adjusting injection targets within their existing treatment. This research addresses a critical gap in managing synkinesis, where current treatments are limited, and could lead to refined protocols that enhance patient quality of life by reducing symptoms and improving facial symmetry. The potential benefits-improved function, aesthetics, and mental well-being-outweigh the minimal risks, as the intervention aligns with established, safe practices.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Current diagnosis of facial synkinesis due to facial nerve paralysis/paresis.
* Scheduled to undergo BT injection for management of facial synkinesis.
* Have undergone > 3 prior BT injection sessions at VUMC for facial synkinesis.
* Able to read and understand English.
* Symptoms of neck tightness, jaw tightness, or headaches.

Exclusion Criteria:

* Cognitive impairment that would preclude the ability to provide informed consent
* Unable to read text on a written survey or computer screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Synkinesis Assessment Questionnaire (SAQ) | Pre-treatment and repeated 5 weeks post-treatment
  This 9-item questionnaire assesses functional status (hyperactive and/or inappropriately active facial muscles) related to facial synkinesis and is already given at each clinic visit as a routine part of clinical practice. The survey is well validated for evaluating synkinesis symptoms in patients with facial nerve injury.
  SAQ scale: 1 = seldom or not at all, 2 = occasionally, or very mildly, 3 = sometimes, or mildly, 4 = most of the time, or moderately, 5 = all the time, or severely
Headache Impact Test (HIT-6) | Pre-treatment and repeated 5 weeks post-treatment
  This 6-item questionnaire seeks to understand the severity of headaches and impact on every-day quality of life. The survey is widely validated for assessing headache symptom and burden. We plan to add in 3 additional questions to this survey including 1) how often do you experience headaches (1 = never or rarely, 2 = 1-2 days a week, 3 = 3-4 days a week, 4 = nearly every day), 2) on a scale of 1-10 (10 = most severe) how severe are your headaches, and 3) I feel as if my Botox injections improved my headaches (Y/N).
  HIT-6 Scale: 1 = Never 2 = Rarely 3 = Sometimes 4 = Very often 5 = Always
Temporomandibular Disorder Questionnare (TMD-7) | Pre-treatment and repeated 5 weeks post-treatment
  This 7-item questionnaire assesses symptoms related to temporomandibular mandibular joint (TMJ) disorder. It asks about jaw pain, tightness, clicking and difficulty eating, among other things. We plan to add in 3 additional questions to this survey including 1) how often do you experience jaw pain/tightness (1 = never or rarely, 2 = 1-2 days a week, 3 = 3-4 days a week, 4 = nearly every day), 2) on a scale of 1-10 (10 = most severe) how severe is your jaw pain/tightness, and 3) I feel as if my Botox injections improved my jaw pain/tightness (Y/N).
  TMD-7 Scale: 1 = Rarely or Never 2 = A few times a month 3 = Once or Twice a Week 4 = Nearly Every Day

CONTACTS AND LOCATIONS:
Overall Officials: Priyesh Patel, MD, Principal Investigator — VUMC

IPD SHARING:
Plan to Share IPD: No